CLINICAL TRIAL: NCT07034365
Title: Risk and Prognosis of Brain Metastasis in Non-Small Cell Lung Cancer: A Multicenter, Prospective, Observational Study
Brief Title: Risk and Prognosis of Brain Metastasis in Non-Small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: LungBM2025
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Brain Metastases From Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC; brain metastases; prognosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples of the patient before and after standardized treatment, as well as baseline tissue samples of intracranial and extracranial lesions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients receiving standard treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This multi-center, prospective, observational study aim to construct a comprehensive model, integrating common clinical pathological parameters, radiographic features and multi-omics data, for assessing the risk and prognosis of brain metastasis in NSCLC. This model is intended to address the following clinical needs: (1) Identify patients at high risk of brain metastasis; (2) Optimize the combined strategies of local and systemic treatments; (3) Predict the survival outcomes of patients with brain metastases from NSCLC and provide evidence-based support for individualized treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer;
* Age≥18 years old;
* KPS score≥70;
* Complete systemic imaging (including brain MRI) before treatment initiation, including contrast-enhanced MRI of the brain;
* Receiving standard treatment;
* Informed consent of the patient.

Exclusion Criteria:

* Multiple primary or metastatic tumors (except early skin cancer, cervical carcinoma in situ that has been treated radically, with no recurrence or progression for more than 5 years);
* Physical examination findings, clinical laboratory abnormalities, or other uncontrolled medical conditions identified by the investigator as potentially interfering with study results interpretation or increasing the patient's risk of - Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are collected all over China, diagnosed with NSCLC.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  The time from enrollment to disease progression or death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.

SECONDARY OUTCOMES:
Intracranial Progression-Free Survival (iPFS) | 2 years
  The time from the enrollment until the documentation of intracranial disease progression or death from any cause. If the patients have extracranial disease progression (without intracranial disease progression), the cutoff date was the date of the first occurrence of extracranial disease progression. Patients who have not progressed at the time of analysis will have their last contact date used as the cutoff date.
Overall Survival (OS) | 2 years
  The time from the start of systemic treatment until death from any cause. Patients who are still alive at the time of analysis will have their last contact date used as the cutoff date.